CLINICAL TRIAL: NCT00498160
Title: Induction of Donor Specific Tolerance in Recipients of Living Kidney Allografts by Donor FCRx Infusion
Brief Title: Induction of Donor Specific Tolerance in Recipients of Live Donor Kidney Allografts by Donor Stem Cell Infusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-7392-041698
Expanded Access: NCT02051673 (No longer available)
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Renal Failure
Keywords: Kidney transplant; Tolerance; Marrow/stem cell transplant
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Living or Deceased Donor Kidney Allograft (Experimental): Recipients with the need for a living kidney allograft are treated with an enriched hematopoetic stem cell infusion from the same living donor. Recipients with the need for a deceased donor kidney allograft are treated with an enriched hematopoetic stem cell infusion from the same deceased donor
  Interventions: Biological: Enriched Hematopoietic Stem Cell Infusion

INTERVENTIONS:
Biological: Enriched Hematopoietic Stem Cell Infusion — Enriched Hematopoietic Stem Cell Infusion

SUMMARY:
The goal of this research study is to establish chimerism and avoid graft-versus-host disease in patients with kidney failure allowing a reduction or cessation of immune-suppressive therapy.

DETAILED DESCRIPTION:
At the present time, kidney transplant recipients must take anti-rejection medication to prevent rejection of the donated kidney. Even with this medication, chronic rejection is the most common cause of late graft loss. The anti-rejection agents themselves are significantly toxic, with side effects including kidney damage, infection and an increased incidence of cancer. The goal of this study is to allow the patient to develop "tolerance" to the transplanted kidney while maintaining a competent immune system. Tolerance enables the transplant recipient's body to recognize the transplanted organ as self rather than foreign tissue. The recipient will not try to reject the donor kidney and the need for anti-rejection medication could be dramatically decreased or eliminated entirely. To accomplish this, patients in this study will receive specially treated bone marrow taken from their kidney donor. Bone marrow transplant has been shown in animal studies and in humans to induce tolerance following organ transplant.

Two factors limit the application of donor marrow transplant to induce tolerance: 1) preparing the patient for transplant (conditioning); and 2) graft-versus-host disease (GVHD). Traditional conditioning destroys the recipient's immune system and requires that the marrow transplant be successful because the patient is unable to fight off infection if the donor cells do not survive. GVHD occurs when donor immune cells recognize the recipient's cells as foreign tissue and attack them. Severe GVHD can result in death. This study utilizes a new approach to conditioning which leaves the patient's immune system intact. The transplant product is depleted of GVHD-producing cells but retains tolerance-promoting facilitating cells, which are intended to ensure the donor and recipient cells coexists peacefully, a state called mixed chimerism. The toxicity of conditioning and transplantation is significantly reduced.

In this study, we will determine the appropriate cell dose to safely establish mixed chimerism following partial conditioning in living donor or deceased donor kidney transplant recipients. The study takes a gradual approach to increasing the cell dose to achieve mixed chimerism. We believe this study will provide a breakthrough in the approach to kidney transplantation. Our goal is to evaluate the potential of safely establishing mixed chimerism to induce tolerance following kidney transplant and reduce or eliminate the need for anti-rejection therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 18 and 65 years and meet the institution's criteria for renal transplantation for end-organ failure
* Patient is receiving first renal transplant
* Patient is receiving a renal transplant only
* The crossmatch is negative between donor and recipient
* Women who are of child bearing potential must have a negative pregnancy test (urine test is acceptable) within 48 hours of initiating total body irradiation (TBI) and agree to use reliable contraception for 1 year following transplant

Note: The subjects do not need to be local residents in order to be eligible for this trial, but must be willing to reside in the area, or within a four hour drive, for the first three months of the protocol so that we can monitor them closely in the early post transplant period. As long as there is insurance or funding that will cover the cost of the transplant and any research related complications, it is not necessary for the subjects to be US citizens to participate in this trial.

Exclusion Criteria:

* Clinically active bacterial, fungal, viral or parasitic infection
* Pregnancy
* Clinical or serologic evidence of viral infection which would preclude the recipient from receiving a kidney transplant
* Previous radiation therapy at a dose which would preclude TBI
* Positive crossmatch between donor and recipient
* Evidence for immunologic memory against donor
* BMI >35 or <18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Level of Donor Chimerism from Enriched Hematopoietic Stem Cell Engraftment | one month to three years
  Tests are done at key time points to monitor for donor chimerism by evaluating presence of bone marrow-derived hematopoietic stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — Talaris Therapeutics Inc.
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Senev A, Tambur AR, Kosmoliaptsis V, Copley HC, Garcia-Sanchez C, Usenko C, Ildstad ST, Leventhal JR. HLA molecular mismatches and induced donor-specific tolerance in combined living donor kidney and hematopoietic stem cell transplantation. Front Immunol. 2024 Mar 27;15:1377535. doi: 10.3389/fimmu.2024.1377535. eCollection 2024. PMID 38601147